CLINICAL TRIAL: NCT03399877
Title: A Study on Accuracy Improvement of Repeated Measure Uroflowmetry- Electromyography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2017-0842
Record Dates: First submitted 2017-12-22; First posted 2018-01-17 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Enuresis
MeSH Terms: conditions — Enuresis

STUDY DESIGN:
Intervention Model Description: Children who meet the inclusion criteria and no exclusion criteria are assigned to perform one of the three test protocols in order of registration according to a computer gererated randomization list. Children who assigned group A perform uroflowmetry-electromyography for the first and subsequently perform uroflowmetry-electromyography again. Children who assigned Group B perform uroflowmetry-electromyography for the first, and subsequently perform sole uroflowmetry. Children who assigned Group C firstly perform sole uroflowmetry and subsequently perform uroflowmetry-electromyography.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combining electromygraphy with uroflowmetry (Active Comparator): Children who assigned group A perform uroflowmetry-electromyography for the first and subsequently perform uroflowmetry-electromyography
  Interventions: Biological: Combining electromyography with uroflowmetry (group A)
- Uroflowmetry (Active Comparator): Children who assigned Group B perform uroflowmetry-electromyography for the first, and subsequently perform uroflowmetry solely.
  Interventions: Biological: Uroflowmetry(Group B)
- Uroflowmetry-Combining electromygraphy with uroflowmetry (Experimental): Children who assigned Group C firstly perform uroflowmetry solely. and subsequently perform uroflowmetry-electromyography.
  Interventions: Biological: Uroflowmetry-Combining electromyography with uroflowmetry (Group C)

INTERVENTIONS:
Biological: Combining electromyography with uroflowmetry (group A) — Children who assigned group A perform uroflowmetry-electromyography for the first and subsequently perform uroflowmetry-electromyography again.
  Arms: Combining electromygraphy with uroflowmetry
Biological: Uroflowmetry(Group B) — Children who assigned Group B perform uroflowmetry-electromyography for the first, and subsequently perform sole uroflowmetry.
  Arms: Uroflowmetry
Biological: Uroflowmetry-Combining electromyography with uroflowmetry (Group C) — Children who assigned Group C firstly perform sole uroflowmetry and subsequently perform uroflowmetry-electromyography.
  Arms: Uroflowmetry-Combining electromygraphy with uroflowmetry

SUMMARY:
Uroflowmetry(UF) has been the standard first-line diagnostic tool for the evaluation of pediatric voiding dysfunction. But recently, UF combined with pelvic flow electromyography(EMG) is emphasized and recommended to analyze the separate contributions of the detrusor and bladder outlet and sole UF is discouraged except for the follow-up study after abnormal UF/EMG result(Bauer et al., 2015). However, electrode itself can disturb pelvic floor relaxation and there is no evidence about necessity of consecutive UF/EMG test. Therefore, the investigators are going to compare three different methods (Primary-Secondary: UF/EMG-UF/EMG, UF/EMG-sole UF, sole UF-UF/EMG)

ELIGIBILITY:
Inclusion Criteria:

1) children aged 5 to 11.9 who visit pediatric urology department for enuresis.

Exclusion Criteria:

1. If children have experience of performing uroflowmetry or uroflowmetry-electromyography.
2. If children do not cooperate on performing the test
3. If enuresis is caused by neurological or anatomical problem.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
maximum flow rate(Qmax=cc/s) | One day
  The maximum flow rate is the most important uroflowmetry index to diagnose bladder outlet obstruction or bladder contractility.

SECONDARY OUTCOMES:
Uroflow curve pattern | One day
  Uroflow curve pattern: There are 5 uroflow curve patterns, bell-shaped, tower-shaped, interrupted-shaped, staccato-shaped and plateau shaped by uroflowmetry. The shape is determined by detrusor contractility and influenced by abdominal straining, coordination with the bladder outlet musculature and any distal anatomic obstruction.
post void residual | One day
  post-void residual(cc): ultrasonographic bladder scan machines calculates bladder volume. PVR measurements in neurologically intact children are highly variable. PVR must be obtained immediately after voiding(<5min)
synergy or dyssynergy between the bladder and the pelvic floor. | One day
  synergy or dyssynergy between the bladder and the pelvic floor is abstained by combining electromyography with uroflowmetry.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology,, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No